CLINICAL TRIAL: NCT00880269
Title: A Phase II Study of Oral Single Agent Panobinostat in Patients With Refractory de Novo or Secondary Acute Myelogenous Leukemia (AML)
Brief Title: Efficacy and Safety of Panobinostat (LBH589) in Patients With Refractory de Novo or Secondary Acute Myelogenous Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2213; 2008-002983-32 (EudraCT Number)
Record Dates: First submitted 2009-03-30; First posted 2009-04-13 (Estimated); Results first posted 2016-09-09 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Refractory Leukemia; Acute Myelogenous Leukemia
Keywords: Acute myeloid leukemia; AML; relapsed acute myeloid leukemia; refractory AML; refractory de novo AML; refractory secondary AML; secondary AML; AML following myelodysplastic syndrome (MDS); AML following antecedent hematological disorder (AHD); AML resistant to therapy
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stratum A (Experimental): patients with refractory acute myelogenous leukemia (AML) initially diagnosed as de novo AML received 60 mg of panobinostat per day on three discontinuous days per week.
  Interventions: Drug: Panobinostat/LBH589
- Stratum B (Experimental): patients with refractory AML initially diagnosed as AML secondary to myelodysplastic syndrome (MDS)/antecedent hematologic disorder (AHD) received 60 mg of panobinostat per day on three discontinuous days per week.
  Interventions: Drug: Panobinostat/LBH589

INTERVENTIONS:
Drug: Panobinostat/LBH589

SUMMARY:
This study was to evaluate the efficacy and safety of single agent oral panobinostat in patients who have refractory de novo or refractory secondary AML.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to study-specific screening procedures
* Life expectancy of ≥ 60 days
* Eastern Cooperative Group (ECOG) performance status ≤ 2
* Refractory AML with confirmed initial diagnosis of de novo AML (excluding APL) - OR- Refractory AML with confirmed initial diagnosis of AML (excluding APL) secondary to AHD or MDS with either condition precedent to AML (MDS/AHD)
* Negative serum pregnancy test (within 7 days of first dose)
* Negative urine pregnancy test immediately prior to first dose

Exclusion Criteria:

* Known HIV
* Psychiatric disorder that interfered with ability to understand the study and give informed consent, and/or would impact study participation or follow-up
* Concurrent use of medications that might prolong the QT interval or of inducing Torsade de Pointes
* Female patients who were pregnant or breast-feeding or patients of childbearing potential who were not willing to use a double barrier method of contraception during the study and for 3 months following the last dose of study drug.
* Male patients whose sexual partner(s) were women of childbearing potential who were not willing to use a double method of contraception, one of which included a condom, during the study and for 3 months after the end of treatment
* Patient unable to swallow capsules
* Patients with impaired gastrointestinal systems which might cause interference with digesting and absorbing panobinostat

Other Protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (38):
- United States (7):
  - University of Chicago Medical Center Dept. of U. of Chicago Hosp(3), Chicago, Illinois
  - Nebraska Methodist Hospital Nebraska Methodist Hospital(2), Omaha, Nebraska
  - North Shore University Hospital North Shore Univ, Manhasset, New York
  - Memorial Sloan Kettering Cancer Center Dept. of MSKCC (2), New York, New York
  - Oregon Health Sciences University Dept. of OHSU (2), Portland, Oregon
  - University of Texas Southwestern Medical Center Dept of Simmons Cancer Center, Dallas, Texas
  - University of Texas/MD Anderson Cancer Center Dept of MD Anderson (14), Houston, Texas
- Australia (6):
  - Novartis Investigative Site, Gosford, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Prahran, Victoria
- Belgium (3):
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Liège
- France (5):
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (3):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Leipzig
- Italy (2):
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Udine, UD
- Novartis Investigative Site, Surquillo, Lima region, Peru
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (2):
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
- Switzerland (2):
  - Novartis Investigative Site, Zurich, Switzerland
  - Novartis Investigative Site, Bern
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Balcova / Izmir
- United Kingdom (4):
  - Novartis Investigative Site, Aberdeen, Scotland
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London

REFERENCES:
- See also: Related Info — http://NovartisClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant flow is based on the full analysis set (FAS) which is the same as the safety set and includes one dose of the study drug.
Pre-assignment Details: Although this study did not complete stage 2, it is considered as a completed study because it follows Simon's optimal two-stage design in each stratum (predefined in the protocol), the study can stop due to futility at the end of Stage 1 and not be considered as a terminated study.
Period: Overall Study
Arm/Group | Stratum A | Stratum B
Started | 32 | 27
Discontinued Treatment | 32 | 27
Completed | 0 | 0
Not Completed | 32 | 27
Not completed — Protocol Violation | 1 | 0
Not completed — Disease Progression | 13 | 11
Not completed — New Cancer Therapy | 1 | 0
Not completed — Death | 4 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Adverse Event | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum A | Stratum B | Total
Number analyzed (Participants) | 32 | 27 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (12.13) | 68.5 (7.75) | 65.5 (10.65)
Gender [Count of Participants; unit: Participants]
  Female | 20 | 8 | 28
  Male | 12 | 19 | 31

OUTCOME MEASURES:

1. Primary Outcome: Best Response as Per Investigator Assessment by Stratum (FAS)
Description: Response to treatment was defined as complete remission rate (CRR). CRR is complete remission (CR) and morphologic CR with incomplete blood count recovery (residual neutropenia or thrombocytopenia) (CRi). To stop or to proceed with Stage 2 of a given stratum of the Simon's optimal 2-stage design was based on the number of patients with CR/CRi and a safety evaluation of the patients from Stage 1 in that stratum. If early results clearly indicated that the drug was not active or worthy of further investigation, enrollment of that particular stratum would be terminated. CR and CRi were assessed by the Investigator according to IWG response Criteria for AML (Cheson et al 2003). As per protocol we would continue to stage II if ≥ 4 patients out of 26 patients enrolled to stage I had a CR or a CRi. As per response observed there was only 1 patient with CR/CRi in stratum A and 2 patients with CR/CRi in Stratum B.
Time Frame: 6 cycles of treatment with a 28-day treatment cycle (Day 168)
Population: Full analysis set (FAS) is the same as the Safety set and includes all patients who received at least one dose of study drug. The FAS was used for final efficacy analyses.
Measure: Number; unit: Percentage of Participants
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 32 | 27
Percentage of Participants
  Complete remission rate (CR/CRi) | 3.1 | 7.4
  Complete remission (CR) | 0 | 3.7
  CR with incomplete blood count recovery (CRi) | 3.1 | 3.7
  Partial remission (PR) | 0 | 0
  Treatment failure | 40.6 | 40.7
  Unknown | 56.3 | 51.9

2. Secondary Outcome: Partial Response Measured in Stratum A and B
Description: As predefined in the study's protocol, stage II was not pursued due to lack of activity (at end of stage I less than 4 patients in each stratum with CR/CRi)
Time Frame: 6 treatment cycles (28-day/treatment cycle)
Population: No secondary analyses were performed since study enrollment was stopped early at stage 1 for lack of evidence of activity.
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Remission Measured in Stratum A and B
Time Frame: 6 treatment cycles (28-day/treatment cycle)
Population: as for outcome 2
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Remission Measured in Stratum A and B
Time Frame: 6 treatment cycles (28-day/treatment cycle)
Population: as for outcome 2
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Event-free Survival Measured in Stratum A and B
Time Frame: 6 treatment cycles (28-day/treatment cycle)
Population: as for outcome 2
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Overall Survival Measured in Stratum A and B
Time Frame: 6 treatment cycles (28-day/treatment cycle)
Population: as for outcome 2
Arm/Group | Stratum A | Stratum B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were followed for 28 days after last dose (Day 467).
Arm/Group | Stratum A | Stratum B
Serious Adverse Events (participants affected / at risk) | 29/32 | 23/27
Other Adverse Events (participants affected / at risk) | 32/32 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum A (N=32) | Stratum B (N=27)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 5
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 8
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 3
Tachycardia (Cardiac disorders) | 0 | 1
Aplasia (Congenital, familial and genetic disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 1 | 2
Fatigue (General disorders) | 3 | 0
General physical health deterioration (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 1
Abdominal infection (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 3
Septic shock (Infections and infestations) | 2 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
General physical condition abnormal (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Systolic hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum A (N=32) | Stratum B (N=27)
Anaemia (Blood and lymphatic system disorders) | 9 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 7
Dry eye (Eye disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 25 | 15
Dry mouth (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 2
Flatulence (Gastrointestinal disorders) | 2 | 0
Gingival bleeding (Gastrointestinal disorders) | 4 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 18 | 14
Odynophagia (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 12 | 8
Asthenia (General disorders) | 4 | 5
Chills (General disorders) | 2 | 0
Fatigue (General disorders) | 10 | 9
Non-cardiac chest pain (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 4 | 3
Pain (General disorders) | 5 | 2
Pyrexia (General disorders) | 16 | 7
Skin infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Blood potassium decreased (Investigations) | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 3
Neutrophil count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 5 | 1
Weight decreased (Investigations) | 4 | 1
White blood cell count decreased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 10 | 9
Dehydration (Metabolism and nutrition disorders) | 4 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 3 | 0
Agitation (Psychiatric disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 5 | 2
Mental status changes (Psychiatric disorders) | 2 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 1
Hypotension (Vascular disorders) | 3 | 3
Thrombophlebitis (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.